CLINICAL TRIAL: NCT00999531
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Multiple Dose Trial to Assess the Safety, Tolerability, and Pharmacokinetics of GS-9411 in Healthy Volunteers
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Multiple Dose Trial of GS-9411 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Thomas O'Riordan, MD, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-221-0107
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Cystic Fibrosis; Mucociliary Clearance; Airway Hydration
Keywords: Cystic Fibrosis; CF; Mucociliary Clearance; Epithelial Sodium Channel Inhibitor; ENaC Inhibitor; Airway Hydration; Amiloride
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): GS-9411 9.6 mg
  Interventions: Drug: GS-9411
- 2 (Experimental): GS-9411 4.8 mg
  Interventions: Drug: GS-9411
- 3 (Experimental): GS-9411 2.4 mg
  Interventions: Drug: GS-9411
- 4 (Placebo Comparator): Saline Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-9411 — Inhaled GS-9411 dissolved in sterile saline
  Arms: 1; 2; 3
Drug: Placebo — Inhaled Placebo, sterile saline
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of repeated doses of GS-9411 in healthy volunteers. GS-9411 is a sodium channel inhibitor, that may restore airway hydration and mucociliary clearance in the lung.

DETAILED DESCRIPTION:
GS-9411 is being evaluated as a potential therapy to improve airway hydration and mucociliary clearance in patients with cystic fibrosis. This study is evaluating the safety and tolerability of 3 dose levels of GS-9411 as an inhaled product, compared to a matched placebo, administered twice daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 65 years of age
* No clinically important abnormal physical findings at Screening
* No clinically relevant abnormalities in the results of laboratory evaluation at Screening
* Must test negative for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) at Screening
* Normal electrocardiogram (ECG) at Screening
* Normal blood pressure (BP) and heart rate (HR) in the absence of any medications for body weight between 50 and 125 kg and within ± 15% of ideal body weight or body mass index (BMI) between 18 and 28 kg/m2 at Screening
* Able to communicate well with the investigator and to comply with the requirements of the entire study
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form
* Nonsmokers of at least 180 days (6 months) duration (< 10 pack/year history) prior to Screening
* Negative for drugs of abuse (including alcohol) at Screening and Day -5
* Must be willing to abstain from alcohol and strenuous exercise during the 48 hours prior to Day -5 and during the study
* Forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted normal for age, gender, and height at Screening and predose
* Normal intraocular pressure (IOP) between 10 and 21 mm Hg at Screening
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g., condoms) during heterosexual intercourse from Day -5 through completion of the study and continuing for at least 90 days from date of last dose of study drug
* Male subjects must refrain from sperm donation from Day -5 through completion of the study and continuing for at least 90 days from the date of last dose of study drug
* Non-lactating females. Females on hormone replacement therapy (estrogen/progesterone) or contraceptive therapy must be stabilized on a product and dose for at least 90 days prior to Screening
* Females must have a negative serum gonadotropin pregnancy test at Screening and Day -1
* Nonpregnant females of childbearing potential must agree to use highly effective (<1% failure rate) contraception during heterosexual intercourse from Screening, throughout the study, and for at least 30 days following the last dose of study drug

Exclusion Criteria:

* Any prior exposure to GS-9411
* Administration of any investigational drug in the period 84 days (12 weeks) prior to Screening; 112 days (16 weeks) if the previous investigational drug was a new chemical entity
* A need for any medication during the period 0 to 5 days prior to Screening, except those deemed by the principal investigator/clinical investigator not to interfere with the outcome of the study
* Existence of any surgical or medical condition which, in the judgment of the clinical investigator, might interfere with the absorption, distribution, metabolism, or excretion of the drug
* Presence or history of allergy requiring treatment. Hay fever is allowed unless it is active or has required treatment within 56 days (8 weeks) of Screening
* Donation or loss of greater than 400 mL of blood in the period 84 days (12 weeks) prior to Screening
* Serious adverse reaction or hypersensitivity to any drug
* Presence or history of any pulmonary diseases (e.g., asthma, emphysema, chronic bronchitis, CF, bronchiectasis)
* Lactating females
* History of glaucoma
* Consumption of drugs and/or herbal preparations capable of inducing hepatic enzyme metabolism (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone, or St. John's Wort) or enzyme-inhibiting agents (e.g., cimetidine) or similar drugs within 28 days (or 5 half-lives of inducing/inhibiting agent, whichever is longer) of Screening
* Major surgery within 180 days (6 months) of the start of this study
* Subjects who have experienced a significant upper or lower respiratory tract infection within the 42 days (6 weeks) prior to Screening
* Subjects with significant history of respiratory, renal, hepatic, cardiovascular (including history of systemic hypertension requiring therapy), metabolic, neurological, hematological, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, may interfere with the study or require treatment which may affect the evaluation of the safety of the study drug
* Subjects with elevated liver enzyme concentrations at Screening and at Day -1
* Hemoglobin level < 130 g/L taken at Screening and at Day -1
* Serum potassium > 5 mEq/L taken at Screening and at Day -1
* Poor venous access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple doses of inhaled GS-9411 in healthy volunteers | 21 Days

SECONDARY OUTCOMES:
Assess the pharmacokinetics of GS-9411 and its metabolites | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hodsman, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network, Ltd., Melbourne, Victoria, Australia

REFERENCES:
- [Derived] O'Riordan TG, Donn KH, Hodsman P, Ansede JH, Newcomb T, Lewis SA, Flitter WD, White VS, Johnson MR, Montgomery AB, Warnock DG, Boucher RC. Acute hyperkalemia associated with inhalation of a potent ENaC antagonist: Phase 1 trial of GS-9411. J Aerosol Med Pulm Drug Deliv. 2014 Jun;27(3):200-8. doi: 10.1089/jamp.2013.1037. Epub 2013 Aug 1. PMID 23905576